CLINICAL TRIAL: NCT05082454
Title: ASCEND - Post Market Clinical Follow-Up Study in Patients Treated With the On-X Ascending Aortic Prosthesis (AAP)
Brief Title: Post Market Clinical Follow-Up Study in Patients Treated With the On-X Ascending Aortic Prosthesis (AAP)
Acronym: ASCEND
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ASCEND
Record Dates: First submitted 2021-09-28; First posted 2021-10-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Disease
Keywords: aortic; valve; stenosis; thoracic; aneurysm; dissection; valved; conduit
MeSH Terms: conditions — Aortic Valve Disease; Constriction, Pathologic; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Open repair — Open repair of the aortic heart valve and ascending thoracic aorta

SUMMARY:
The ASCEND post-market clinical follow-up study is undertaken to evaluate safety and clinical performance of the On-X Ascending Aortic Prosthesis (AAP) used in surgical aortic valve replacement.

DETAILED DESCRIPTION:
In this study patients will be observed that receive an On-X AAP implant for the treatment of a diseased, damaged, or malfunctioning native or prosthetic heart valve. The On-X AAP will be implanted at the discretion of the treating physician. Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with the On-X AAP. Written informed consent, specifically allowing the use of clinical records for this observational study, will be obtained from every patient in Europe and every patient that is alive in the US prior to data collection where required. In Europe, every patient will be enrolled prospectively prior to the intervention.

In the US, patients can be enrolled retrospectively after the intervention or prospectively prior to the intervention. The data from patients who have died following their implant will be recorded in the database without the requirement for written informed consent after IRB approval.

The period of data collection will be approximately 60 + 6 months (depending on the date of the last follow-up visit) from the surgery for each patient.

Echocardiography images at prior to discharge, at 12 months, 60 months will be evaluated by a CoreLab. All adverse events defined in the Clinical Event Committee (CEC) charter will be adjudicated by the CEC.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at time of On-X AAP implant
* Patient understands and has signed the Informed Consent Form:

  * Prior to implant of On-X AAP or
  * Post implant (US only) or
  * Patient died prior to enrollment (US only)
* Patient is willing and able to participate in follow-up

Exclusion Criteria:

* Patient unable to tolerate anticoagulation therapy
* Patient with active endocarditis at the time of his / her On-X AAP implant
* Patient participates / participated in another clinical investigation which may interfere / may have interfered with the effectiveness of anticoagulation therapy
* Patient has anomalous anatomy or medical, surgical, psychological or social history or conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results
* Patients in which On-X AAP is implanted in combination with AMDS or FET
* Patient's life expectancy is less than 3 years in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients (≥ 18 years of age) who either underwent (US only) or will be undergoing (Europe and US) implant of the On-X AAP for aortic valve and ascending aorta replacement and who meet the criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | at discharge to home or to rehabilitation
  Rate of in-house all-cause mortality

SECONDARY OUTCOMES:
All-cause Mortality | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of all-cause mortality
Valve-related mortality | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of valve-related mortality
Reoperation | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with reoperation
Explant | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with explant of On-X AAP (including heart valve)
Endocarditis | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with endocarditis
Embolism | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with embolism
Thromboembolism | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with peripheral thromboembolism
Bleeding | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with major bleeding
Transient ischemic attack | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with transient ischemic attack (TIA)
Stroke | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with new stroke (ischemic and hemorrhagic) (mRS > mRS at baseline)
Ischemic stroke | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with new ischemic stroke (mRS > mRS at baseline)
Hemorrhagic stroke | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with new hemorrhagic stroke (mRS > mRS at baseline)
Valve deterioration | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with structural valve deterioration
Non-structural dysfunction | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with non-structural dysfunction
Valve thrombosis | 30-day, 1 year, 2 years, 3 years, 4 years, 5 years
  Rate of patients with valve thrombosis
NYHA | 1 year, 3 years, 5 years
  NYHA Functional Class

CONTACTS AND LOCATIONS:
Overall Officials: Davide Pacini, Prof. Dr., Principal Investigator — Policlinico S. Orsola-Malpighi
Locations (11):
- United States (3):
  - Geisinger Health System, Danville, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - VCU Medical Center Main Hospital, Richmond, Virginia
- Germany (2):
  - Medizinische Hochschule Hannover (MHH), Hanover
  - University Hospital Magdeburg, Magdeburg
- Policlinico S. Orsola-Malpighi, Bologna, Italy
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- United Kingdom (3):
  - Castle Hill Hospital, Cottingham
  - St Bartholomew's Hospital, London
  - Newcastle Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No